CLINICAL TRIAL: NCT06215846
Title: Phase I Clinical Study on the Safety, Tolerability, and Pharmacokinetics of Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001) in Patients With Malignant Solid Tumors
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of BioTTT001 in Patients With Malignant Solid Tumors
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Bio-Targeting Therapeutics Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCT-01-101
Record Dates: First submitted 2023-11-27; First posted 2024-01-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor
Keywords: Oncolytic virus; IL-12; Adenovirus
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioTTT001 injection (Experimental): BioTTT001 is administered as a single Intratumoral injection. The dose groups to be infusion were 5×10^9 viral particle (VP) ,5×10^10 VP and 5×10^11 VP based on the 3+3 dose escalation principle.
  Interventions: Biological: BioTTT001 injection

INTERVENTIONS:
Biological: BioTTT001 injection — BioTTT001 is administered as a single Intratumoral injection. The dose groups to be infusion were 5×10^9 VP, 5×10^10 VP and 5×10^11 VP based on the 3+3 dose escalation principle.

SUMMARY:
This is a Phase 1 open-label study to evaluate the safety, tolerability, and pharmacokinetics of Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001) at dose of 5×10∧9VP、5×10∧10VP、5×10∧11VP in Patients With Malignant Solid Tumors. Subjects will be treated with a single dose of BioTTT001 Injection after the screening period.

DETAILED DESCRIPTION:
This study is a single arm, open label, single center dose escalation trial. Three study drug dosage groups are pre-set, namely 5 × 10∧9VP、5 × 10∧10VP、 5 × 10∧11VP. According to the principle of dose escalation from low to high, the "3+3" dose escalation method is adopted. In theory, in order to protect the safety of the subjects, during the DLT observation phase of the same dose group, the first subject in each dose group can only be enrolled in the second subject after at least 2 weeks after administration. The DLT observation period for each subject is 28 days after the first administration, and the last subject in each dose group can only enter the next dose escalation after completing the DLT observation period. At least 3 subjects are enrolled in each dose group, and each subject only receives one corresponding dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 80 years old (including the threshold), no gender restrictions.
2. Patients with histologically and/or cytologically confirmed malignant solid tumors, who have experienced at least one-line standard treatment failure or intolerance, or lack standard treatment options. Focus on malignancies in the head and neck, colorectal cancer, skin malignancies, and cervical cancer.
3. At least one assessable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
4. Assessed by the investigators to have lesions suitable for intratumoral injection (assessable lesions and intratumoral injection lesions can refer to the same lesion).

Exclusion Criteria:

1. Known allergy to the investigational drug or its components.
2. Previous treatment with other adenovirus drugs.
3. Patients with active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, etc.), except type 1 diabetes, hypothyroidism that only needs hormone replacement therapy, and skin diseases that do not need systemic treatment (such as vitiligo, psoriasis or alopecia).
4. Patients who have not recovered from the adverse reactions of previous treatments (the treatment-related toxicity ≤ grade 2, except for alopecia, pigmentation or other tolerable events judged by the investigator ).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 28 days within BioTTT001 injection
  The incidence and severity of all types of adverse events evaluated based on NCI-CTCAE V5.0 assessment
MTD | 28 days within BioTTT001 injection
  Maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Plasma Adenovirus (ADV) copies | 28 days within BioTTT001 injection
  Pharmacokinetic Study (PK): Copies of ADV in plasma at various sampling points.
ADV copies in various sites | 28 days within BioTTT001 injection
  Viral Shedding Analysis: Copies of ADV in swabs of injection sites, rectal swabs, throat swabs, and urine samples at various sampling points.
Serum interleukin-12 (IL-12) level | 28 days within BioTTT001 injection
  Expression levels of IL-12 at various sampling points in serum.
Serum neutralizing antibody level | 28 days within BioTTT001 injection
  Immunogenicity assessment through neutralizing antibody detection.
ORR | From date of the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Objective response rate (ORR) as assessed by the investigators.
DCR | From date of the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Disease control rate (DCR) as assessed by the investigators.
PFS | From date of the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression-free survival (PFS) as assessed by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenning Wang, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy; Funan Liu, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy
Locations (1):
- The First Affiliated Hospital of China Medical Univeristy, Shenyang, Liaoning, China